CLINICAL TRIAL: NCT03477916
Title: Fecal Microbial Transplantation and Fiber Supplementation in Participants With Obesity and Metabolic Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: W. Garfield Weston Foundation (Unknown)
Responsible Party: Principal Investigator, Karen Madsen, Director, CEGIIR Professor, Division of Gastroenterology, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00076642
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo FMT and cellulose) (Other)
  Interventions: Biological: Placebo FMT; Dietary Supplement: Cellulose
- FMT only (FMT followed by cellulose) (Experimental)
  Interventions: Biological: FMT; Dietary Supplement: Cellulose
- Prebiotic only (Placebo FMT and prebiotic fiber) (Other)
  Interventions: Biological: Placebo FMT; Dietary Supplement: Prebiotic Fiber
- FMT + prebiotic fiber (Experimental)
  Interventions: Biological: FMT; Dietary Supplement: Prebiotic Fiber

INTERVENTIONS:
Biological: FMT — fecal microbial transplantation (FMT)
  Arms: FMT + prebiotic fiber; FMT only (FMT followed by cellulose)
Biological: Placebo FMT — Placebo fecal microbial transplantation (FMT)
  Arms: Control (Placebo FMT and cellulose); Prebiotic only (Placebo FMT and prebiotic fiber)
Dietary Supplement: Prebiotic Fiber — combined fiber supplement of resistant starch type 4, acacia gum, and soluble corn fiber
  Arms: FMT + prebiotic fiber; Prebiotic only (Placebo FMT and prebiotic fiber)
Dietary Supplement: Cellulose — Cellulose
  Arms: Control (Placebo FMT and cellulose); FMT only (FMT followed by cellulose)

SUMMARY:
Obesity is increasing in western society at a rapid rate and is associated with metabolic and cardiovascular disease. Although genetics, improper diet, and sedentary lifestyle are known to be factors that can cause obesity, there is a new idea that certain gut microbes may also be involved. Patients who are obese tend to have different kinds of gut microbes compared with lean healthy individuals. Previous studies have shown that changing the gut microbes of obese individuals by doing a fecal transplant (FMT) using gut microbes from a lean individual improves insulin resistance. However, the effects were not maintained. In addition, research has highlighted a necessary role for dietary fiber in the maintenance of microbes required for human health and also that increasing dietary fiber can reduce inflammation that is associated with insulin resistance. This project builds on the findings that gut microbes can be modulated by both FMT and dietary fiber supplementation and will examine if combining these two treatments can increase the effectiveness of these treatments.

The objective of this study is to use fecal microbial transplant to change the gut microbes of obese individuals to those seen in lean individuals and then to use fiber supplements to help maintain the beneficial effects. In this study, overweight individuals who have metabolic syndrome will receive a fecal transplant using a pill form and then consume a variety of fiber supplements for 6 weeks. Effects on metabolic parameters, quality of life, weight, and dietary intake will be followed. Microbial composition will be measured in stool samples.

DETAILED DESCRIPTION:
Phase: This is a phase II clinical trial.

Methodology: This is an exploratory, four-arm, parallel design, randomized placebo-controlled intervention study.

Study Duration: 12 weeks Study Center(s): This is a single center trial at the University of Alberta

Objectives:The objective of this study is to determine if fecal microbial transplantation (FMT) combined with supplementation with a combined fiber supplement of resistant starch type 4, acacia gum, and soluble corn fiber has a clinically significant effect on metabolic outcomes in obese subjects with metabolic syndrome

Primary Outcome: Changes in insulin sensitivity between the time of screening and 6 weeks following treatment.

Secondary Outcomes:

* Changes in Body weight and anthropometric parameters between baseline and week 6.
* Changes in HbA1C, fasting glucose, glucose tolerance test between baseline and week 6
* Changes in fasting lipid profile between baseline and week 6
* Changes in blood pressure between baseline and week 6
* Quality of life and satiety between baseline and week 6
* Changes in serum levels of leptin, adiponectin, ghrelin, CRP, TNF-α, IL-6, LPS, LPS-binding protein and zonulin between baseline and week 6
* Changes in stool microbiota composition between baseline and week 6
* Changes in stool short chain fatty acid composition between baseline and week 6

Number of Subjects: 68

Diagnosis and Main Inclusion Criteria

Primary Diagnosis:

• BMI > 30

Key Inclusion Criteria:

* Age 18-64 years at screening
* Total body weight fluctuation over the last 6 months <10%
* Fasting plasma glucose > 5.6 mmol/L OR HgbA1c ≥6.5% (with or without taking an oral antidiabetic medication)
* At least one of the following:

  * Fasting triglyceride ≥1.7 mmol/L (with or without taking a statin or fibrate)
  * HDL cholesterol <1.03 mmol/L in males or <1.29 mmol/L in females (with or without taking a statin or fibrate)
  * Known diagnosis of hypertension OR systolic blood pressure ≥130 or diastolic blood pressure ≥85 mmHg (with or without taking at least one antihypertensive agent).

Study Product, Dose, Route, Regimen FMT:

* 50 gm of screened and encapsulated single donor stool (approximately 20-30 capsules) taken by mouth on day 1 of the trial after having fasted overnight and completed a bowel prep with Pico-Salax®.
* Placebo pills will contain microcrystalline cellulose

Soluble corn fiber (PROMITOR®: Tate&Lyle)

* Women: 4.5 gm of PROMITOR by mouth days 1-3 increased to 9 gm daily from day 4 until trial completion.
* Men: 5.5 gm of PROMITOR by mouth days 1-3 increased to 11 gm by mouth daily from day 4 until trial completion.

Resistant Wheat Starch 4 (Fibersym®: MGP Ingredients):

* Women: 4.5 gm of powdered RS4 by mouth days 1-3 increased to 9 gm by mouth daily from day 4 until trial completion.
* Men: 5.5gm of powdered RS4 by mouth days 1-3 increased to 11 gm by mouth daily from day 4 until trial completion.

Acacia Gum (Pre-Hydrated Gum Arabic: TIC GUMS):

* Women: 4.5 gm of powdered acacia gum by mouth days 1-3 increased to 9 gm by mouth daily from day 4 until trial completion.
* Men: 5.5gm of powdered acacia gum by mouth days 1-3 increased to 11 gr by mouth daily from day 4 until trial completion.

Duration of administration:

FMT: Single dose of 50gm donor stool or placebo (microcrystalline cellulose) on day 1.

Fiber: Daily administration until completion at week 6

Reference therapy Both FMT and Fiber will be placebo matched as reference therapy.

Statistical Methodology: Study groups with by analyzed by pair-wise comparison with evaluation of means between and across groups using paired or unpaired t-tests for continuous outcomes and chi-squared tests for dichotomous ones. Multivariable predictors of change in relevant outcomes will be identified using appropriately constructed and calibrated linear regression models for continuous outcomes or logistic regression models for dichotomous ones.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 and < 65 years at the time of screening

  * BMI > 30
  * Total body weight fluctuation over the last 6 months less than 10%
  * Fasting plasma glucose (FPG): 1) > 5.6 mmol/L OR Hemoglobin A1c ≥6.5% (with or without taking an oral antidiabetic medication).
  * At least one of the following criterion:

    1. Fasting triglyceride ≥1.7 (TG) mmol/L (with or without taking a statin or fibrate)
    2. HDL cholesterol <1.03 mmol/L in males or <1.29 mmol/L in females (with or without taking a statin or fibrate)
    3. Established diagnosis of hypertension OR SBP ≥130 or DBP ≥85 mmHg (with or without taking at least one antihypertensive agent).

Exclusion Criteria:

* • Systolic blood pressure ≥180 or diastolic blood pressure ≥110 mmHg at screening.

  * Triglyceride ≥6 mmol/L.
  * Acute infectious or inflammatory condition over the presiding 4 weeks.
  * Current or recent use (Previous 6 months) of insulin for diabetes control.
  * History of oropharyngeal or significant esophageal dysphagia, inflammatory bowel disease, colon cancer, or colonic polyps with high grade dysplasia.
  * History of autoimmune conditions or chronic inflammatory condition, such as rheumatoid arthritis, chronic active hepatitis B or C, HIV, chronic pancreatitis, advanced NASH, or liver cirrhosis.
  * Active malignancy.
  * Active substance abuse or excessive EtOH (defined as >2 X 8oz drinks/d).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | Change between the time of screening and 6 weeks following treatment.
  The primary endpoint is the change in insulin sensitivity between the time of screening and 6 weeks following treatment.

SECONDARY OUTCOMES:
BMI | Changes between baseline and 6 and 12 weeks
  weight and height will be combined to report changes in BMI in kg/m^2 between baseline and 6 and 12 weeks
Waist to hip circumferences | Changes between baseline and 6 and 12 weeks
  Changes in waist to hip circumferences between baseline and 6 and 12 weeks
HbA1C | Changes between baseline and 6 and 12 weeks
  Changes HbA1C between baseline and 6 and 12 weeks
fasting glucose | Changes between baseline and 6 and 12 weeks
  Changes fasting glucose between baseline and 6 and 12 weeks
oral glucose tolerance | Changes between baseline and 6 and 12 weeks
  Changes in oral glucose tolerance between baseline and 6 and 12 weeks
Fasting lipid profile | Changes between baseline and 6 and 12 weeks
  Changes in Fasting lipid profile between baseline and 6 and 12 weeks
blood pressure | Changes between baseline and 6 and 12 weeks
  Changes in blood pressure between baseline and 6 and 12 weeks
EuroQol five dimensions questionnaire (EQ-5D™) | Changes between baseline and 6 and 12 weeks
  Changes in EuroQol five dimensions questionnaire scores to arrive at the participants quality of life between baseline and 6 and 12 weeks
SLIM Hunger and Satiety Questionnaire | Changes between baseline and 6 and 12 weeks
  The SLIM Hunger and satiety questionnaire scores used to arrive at the participants feelings of hunger and satiety. Changes in reported feelings of Hunger and Satiety between baseline and 6 and 12 weeks
serum levels of leptin, adiponectin, ghrelin, CRP, TNF-α, IL-6, LPS, and LPS-binding protein | Changes between baseline and 6 and 12 weeks
  Changes in serum levels of leptin, adiponectin, ghrelin, CRP, TNF-α, IL-6, LPS, and LPS-binding protein between baseline and 6 and 12 weeks
fecal microbiota composition | Changes between baseline and 6 and 12 weeks
  Changes in fecal microbiota composition between baseline and 6 and 12 weeks
stool short chain fatty acid composition | Changes between baseline and 6 and 12 weeks
  Changes in stool short chain fatty acid composition between baseline and 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Madsen, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mocanu V, Zhang Z, Deehan EC, Kao DH, Hotte N, Karmali S, Birch DW, Samarasinghe KK, Walter J, Madsen KL. Fecal microbial transplantation and fiber supplementation in patients with severe obesity and metabolic syndrome: a randomized double-blind, placebo-controlled phase 2 trial. Nat Med. 2021 Jul;27(7):1272-1279. doi: 10.1038/s41591-021-01399-2. Epub 2021 Jul 5. PMID 34226737